CLINICAL TRIAL: NCT05478226
Title: ADAMTSL4 in Idiopathic Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension
Brief Title: ADAMTSL4 in Idiopathic Pulmonary Hypertension and CTEPH
Status: Completed | Type: Observational
Sponsor: Wei Huang (Other)
Responsible Party: Sponsor-Investigator, Wei Huang, Professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2019XMSB000726
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control group: healthy people as control group
- IPAH group: patients with IPAH as IPAH group
  Interventions: Other: drugs or BPA
- CTEPH group: patients with CTEPH as CTEPH group
  Interventions: Other: drugs or BPA
- group D: Including CTEPH group and IPAH group
  Interventions: Other: drugs or BPA

INTERVENTIONS:
Other: drugs or BPA — PAH target drugs，for example， Tadanafiland, Maxitensin, Prostacyclins, riociguat and etc. CTEPH treat with balloon pulmonary angioplasty or riociguat
  Groups: CTEPH group; IPAH group; group D

SUMMARY:
ADAMTSL4 (A disintegrin and metalloproteinase with thrombospondin motifs like) is a member of the ADAMTSL family. ADAMTSL4 is one of the family of 7 ADAMTS-Like proteins, themselves part of the Thrombospondin type 1 repeat (TSR) superfamily of proteins. These 7 proteins are divided into two distinct clades, of which ADAMTSL4 and ADAMTS-Like 6 form part of one clade, differing from ADAMTS-Like 1, ADAMTS-Like 3 and ADAMTS-Like 7 by lacking immunoglobulin repeat regions. ADAMTSL4 is widely expressed in brain, colon, heart, kidney, liver, lung, pancreas and spleen, yet, its precise role is unclear. in addition, ADAMTSL4 protein high expression to the medial layer of the arterial wall, and medial vascular smooth muscle cells specifically.

DETAILED DESCRIPTION:
The objectives of the present study aimed to confirm ADAMTSL4 levels in the proteomics between healthy control population and patients with IPAH，to analyze the expression levels of ADAMTSL4 between patients with IPAH and CTEPH, and to investigate whether serum levels of ADAMTSL4 might be used as biomarkers of disease severity in these patient populations.

ELIGIBILITY:
Inclusion Criteria:

- Healthy people，patients with IPAH，patients with CTEPH

Exclusion Criteria:

- tumour，infection，Pregnancy, suckling period， Mental disorders，

Other types of PAH except CTEPH and IPAH

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with IPAH and CTEPH compliance with 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Association of clinic index and ADAMTSL4 expression level | 2018-2022
  The expression and its clinical relevance of ADAMTSL4 expression level in plasma or pulmonary tissue in patients with IPAH and CTEPH

CONTACTS AND LOCATIONS:
Overall Officials: Wei Huang, Phd, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the First Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The IPD is undecided